CLINICAL TRIAL: NCT01410474
Title: A Phase 3, Multicenter, Open-label Study to Evaluate Immunogenicity and Safety of Novartis Meningococcal ACWY Conjugate Vaccine (MenACWY-CRM) in Healthy Subjects From 2 to 18 Years in Taiwan
Brief Title: Immunogenicity and Safety of Meningococcal ACWY Conjugate Vaccine in Healthy Subjects From 2 to 18 Years in Taiwan
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Collaborators: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V59_49
Record Dates: First submitted 2011-08-03; First posted 2011-08-05 (Estimated); Results first posted 2014-09-22 (Estimated); Last update posted 2014-09-22 (Estimated); Status verified 2014-09

CONDITIONS: Bacterial Meningitis
Keywords: Meningococcal; ACWY; bacterial meningitis; conjugate vaccine; healthy; children; adolescents; Taiwan
MeSH Terms: conditions — Meningitis, Bacterial

ARMS (1):
- 2-18 years (Experimental)
  Interventions: Biological: Meningococcal ACWY conjugate vaccine

INTERVENTIONS:
Biological: Meningococcal ACWY conjugate vaccine — All subjects received a single dose of Meningococcal ACWY conjugate vaccine and had blood draw at day 1 and day 29.

SUMMARY:
This study will evaluate the immunogenicity and safety of a single injection of Novartis Meningococcal ACWY conjugate vaccine in healthy subjects from 2 to 18 years in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects from 2 up to and including 18 years of age
2. Who are in good health as determined by : medical history, physical exam,clinical judgment of the investigator, who have a negative urine pregnancy test for female subjects ≥11 years of age

Exclusion Criteria:

Individuals not eligible to be enrolled in the study were those:

1. Who had a previous confirmed or suspected disease caused by N. meningitidis.
2. Who had household contact with and/or intimate exposure to an individual with culture-proven N. meningitidis infection within 60 days prior to enrolment.
3. Who have previously been immunized with a meningococcal vaccine or vaccine containing meningococcal antigen(s) (licensed or investigational).
4. Who have received any vaccines within 14 days (for inactivated vaccines) or 28 days (for live vaccines) prior to enrolment in this study or who are planning to receive any vaccine within 30 days from the study vaccines.
5. Who have experienced within the 7 days prior to enrolment significant acute infection or have experienced fever within 3 days prior to enrolment.
6. Who have any serious acute, chronic or progressive who have epilepsy or any progressive neurological disease or history of Guillain-Barre syndrome.
7. Who have a history of any anaphylaxis, serious vaccine reactions, or allergy to any vaccine components.
8. Who have a known or suspected impairment/alteration of immune function, either congenital or acquired
9. Who are known to have a bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
10. Who have Down's syndrome or other known cytogenic disorders.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 341 (Actual)
Dates: Start 2011-08; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Li Min Huang, Dr., Principal Investigator — Dr. Li Min Huang, National Taiwan University Hospital; Nan Chang Chiu, Dr., Principal Investigator — Mackay Memorial Hospital; Shu Jen Yeh, Dr., Principal Investigator — Far Eastern Memorial Hospital
Locations (3):
- China (3):
  - Mackay Memorial Hospital,, Taipei, Taiwan
  - National Taiwan University Hospital, Taipei, Taiwan
  - Far Eastern Memorial Hospital,, Taipei, Taiwan

REFERENCES:
- [Derived] Huang LM, Chiu NC, Yeh SJ, Bhusal C, Arora AK. Immunogenicity and safety of a single dose of a CRM-conjugated meningococcal ACWY vaccine in children and adolescents aged 2-18 years in Taiwan: results of an open label study. Vaccine. 2014 Sep 8;32(40):5177-84. doi: 10.1016/j.vaccine.2014.07.063. Epub 2014 Jul 27. PMID 25075804

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled at three study centres in Taiwan.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- 2-10 Years: Subjects 2-10 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1.
- 11-18 Years: Subjects 11-18 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1.
Period: Overall Study
Arm/Group | 2-10 Years | 11-18 Years
Started | 173 | 168
Completed | 173 | 167
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was done on all the enrolled subjects.
Groups:
- Total: Total of all reporting groups
Arm/Group | 2-10 Years | 11-18 Years | Total
Number analyzed (Participants) | 173 | 168 | 341
Age, Continuous [Mean (Standard Deviation); unit: Years] | 6.3 (2.6) | 14.0 (2.2) | 10.1 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 88 | 180
  Male | 81 | 80 | 161

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Overall Subjects With Seroresponse, Directed Against Neisseria Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as the percentage of subjects with hSBA seroresponse and associated 95% Clopper-Pearson confidence interval (CI), directed against N. meningitidis serogroups A, C, W and Y, evaluated by serum bactericidal assay using human complement (hSBA), at 28 days after one vaccination of MenACWY-CRM (day 29).
  Seroresponse is defined as:
  1. for subjects with a prevaccination hSBA titer <1:4, a postvaccination hSBA titer ≥1:8.
  2. for subjects with a prevaccination hSBA titer ≥1:4, an increase in hSBA titer of at least four times the prevaccination titer.
Time Frame: Day 1 and Day 29
Population: Analysis was done on modified intention-to-treat (MITT) population i.e subjects in the exposed population who provided evaluable serum samples whose assay results were available for at least one serogroup on day 1 and/or day 29.
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Groups:
- Overall (2 to 18 Years): Subjects 2 to 18 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1.
Arm/Group | Overall (2 to 18 Years)
Number analyzed (Participants) | 336
Percentages of Subjects
  MenA (N=335) | 83 [79 to 87]
  MenC (N=333) | 93 [90 to 96]
  MenW (N=334) | 50 [45 to 55]
  MenY (N=333) | 65 [60 to 70]

2. Secondary Outcome: Percentage of Subjects With Seroresponse, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination, by Age Group
Description: Immunogenicity was measured as the percentage of subjects with hSBA response and associated 95% CI, directed against N. meningitidis serogroups A, C, W and Y, at Day 29, by age groups.
  Seroresponse is defined as:
  1. for subjects with a prevaccination hSBA titer <1:4, a postvaccination hSBA titer ≥1:8.
  2. for subjects with a prevaccination hSBA titer ≥1:4, an increase in hSBA titer of at least four times the prevaccination titer.
Time Frame: Day 1 and Day 29
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2-10 Years | 11-18 Years
Number analyzed (Participants) | 170 | 166
Percentages of Subjects
  Men A (N=170,165) | 77 [70 to 83] | 89 [83 to 93]
  MenC (N=167,166) | 92 [86 to 95] | 95 [90 to 97]
  MenW (N=168,166) | 54 [46 to 62] | 46 [38 to 54]
  MenY (N=167,166) | 61 [53 to 69] | 69 [62 to 76]

3. Secondary Outcome: Geometric Mean Titers (GMTs) of Subjects, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as hSBA GMTs and associated 95% CI, against N. meningitidis serogroups A, C, W and Y, before the vaccination (Day 1) and 28 days after MenACWY-CRM vaccination (Day 29), by age group and overall.
Time Frame: Day 1 and 29
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: hSBA Titers
Arm/Group | 2-10 Years | 11-18 Years | Overall (2 to 18 Years)
Number analyzed (Participants) | 170 | 166 | 336
hSBA Titers
  MenA at Day 1(N=170,165,335) | 2.05 [1.92 to 2.2] | 2.2 [2.05 to 2.36] | 2.12 [2.02 to 2.24]
  MenA at Day 29(N=170,165,335) | 32 [24 to 43] | 88 [66 to 117] | 53 [42 to 65]
  MenC at Day 1 (N=167,166,333) | 2.66 [2.35 to 3.02] | 3.64 [3.21 to 4.12] | 3.11 [2.83 to 3.42]
  MenC at Day 29 (N=167,166,333) | 117 [93 to 147] | 273 [218 to 342] | 179 [151 to 211]
  MenW at Day 1 (N=168,166,334) | 7.32 [5.65 to 9.49] | 15 [12 to 19] | 10 [8.62 to 13]
  MenW at Day 29 (N=168,166,334) | 49 [40 to 60] | 104 [85 to 127] | 71 [61 to 82]
  MenY at Day 1 (N=167,166,333) | 3.21 [2.69 to 3.83] | 3.95 [3.31 to 4.71] | 3.56 [3.12 to 4.06]
  MenY at Day 29 (N=167,166,333) | 26 [20 to 33] | 56 [43 to 72] | 38 [31 to 46]

4. Secondary Outcome: Geometric Mean Ratios (GMRs) of Subjects, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as ratio of postvaccination GMTs to prevaccination GMTs and associated 95% CI, against N. meningitidis serogroups A, C, W and Y, at 28 days after MenACWY-CRM vaccination (Day 29), by age group and overall.
Time Frame: Day 1 and Day 29
Population: Analysis was done on MITT population
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | 2-10 Years | 11-18 Years | Overall (2 to 18 Years)
Number analyzed (Participants) | 170 | 166 | 336
Ratio
  MenA(N=170,165,335) | 16 [12 to 21] | 40 [30 to 53] | 25 [20 to 31]
  MenC (N=167,166,333) | 44 [35 to 56] | 75 [59 to 95] | 57 [48 to 69]
  MenW (N=168,166,334) | 6.66 [5.19 to 8.54] | 6.91 [5.39 to 8.85] | 6.78 [5.63 to 8.16]
  MenY (N=167,166,333) | 8.02 [6.09 to 11] | 14 [11 to 19] | 11 [8.67 to 13]

5. Secondary Outcome: Percentage of Subjects With hSBA Titer ≥1:8, Directed Against N. Meningitidis Serogroups A, C, W and Y After MenACWY-CRM Vaccination
Description: Immunogenicity was measured as the percentage of subjects with hSBA titer ≥1:8 and associated 95% CI, before vaccination (Day 1) and 28 days after MenACWY-CRM vaccination (Day 29), bye age group and overall.
Time Frame: Day 1 and 29
Population: Analysis was done on MITT population
Measure: Number (95% Confidence Interval); unit: Percentages of Subjects
Arm/Group | 2-10 Years | 11-18 Years | Overall (2 to 18 Years)
Number analyzed (Participants) | 170 | 166 | 336
Percentages of Subjects
  MenA at Day 1 (N=170,165,335) | 1 [0 to 4] | 4 [2 to 9] | 3 [1 to 5]
  MenA at Day 29 (N=170,165,335) | 77 [70 to 83] | 90 [84 to 94] | 83 [79 to 87]
  MenC at Day 1 (N=167,166,333) | 11 [7 to 17] | 23 [17 to 31] | 17 [13 to 22]
  MenC at Day 29 (N=167,166,333) | 95 [90 to 98] | 98 [95 to 100] | 96 [94 to 98]
  MenW at Day 1 (N=168,166,334) | 47 [39 to 55] | 70 [62 to 77] | 58 [53 to 64]
  MenW at Day 29 (N=168,166,334) | 93 [88 to 96] | 99 [96 to 100] | 96 [93 to 98]
  MenY at Day 1 (N=167,166,333) | 22 [16 to 29] | 26 [19 to 33] | 24 [19 to 29]
  MenY at Day 29 (N=167,166,333) | 78 [71 to 84] | 86 [79 to 91] | 82 [77 to 86]

6. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic Adverse Events After MenACWY-CRM Vaccination, Age 2 to 5 Years
Description: Safety was assessed as the number of subjects aged 2 to 5 years who reported solicited local and systemic adverse events (AEs) within days 1 through 7 after MenACWY-CRM vaccination.
Time Frame: From day 1 through day 7 postvaccination
Population: Analysis was done on safety population i.e. the subjects in the exposed population who provided post-baseline safety data.
Measure: Number; unit: Subjects
Groups:
- 2-5 Years: Subjects 2-5 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1
Arm/Group | 2-5 Years
Number analyzed (Participants) | 72
Subjects
  Injection site tenderness | 27
  Injection site erythema | 7
  Injection site induration | 6
  Change in eating habits | 2
  Sleepiness | 3
  Irritability | 5
  Vomiting | 7
  Diarrhea | 2
  Rash - Any | 4
  Rash - Urticarial | 1
  Fever (≥38°C) | 4

7. Secondary Outcome: Number of Subjects Who Reported Solicited Local and Systemic AEs After MenACWY-CRM Vaccination, Age 6 to 18 Years
Description: Safety was assessed as the number of subjects aged 6 to 18 years who reported solicited local and systemic AEs within days 1 through 7 after MenACWY-CRM vaccination.
Time Frame: From day 1 through day 7 postvaccination
Population: Analysis was done on safety population.
Measure: Number; unit: Subjects
Groups:
- 6-10 Years: Subjects 6-10 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1
- Overall (6-18 Years): Subjects 6-18 years of age received one 0.5 mL dose of MenACWY-CRM vaccination as intramuscular (IM) injection at Day 1
Arm/Group | 6-10 Years | 11-18 Years | Overall (6-18 Years)
Number analyzed (Participants) | 101 | 167 | 268
Subjects
  Injection site pain | 37 | 62 | 99
  Injection site erythema | 17 | 17 | 34
  Injection site induration | 14 | 12 | 26
  Chills | 2 | 6 | 8
  Nausea | 10 | 10 | 20
  Malaise | 13 | 35 | 48
  Myalgia | 20 | 49 | 69
  Arthralgia | 3 | 13 | 16
  Headache | 11 | 29 | 40
  Rash - Any | 7 | 4 | 11
  Rash - Urticarial | 3 | 3 | 6
  Fever (≥38°C) | 3 | 2 | 5

ADVERSE EVENTS:
Time Frame: Throughout the study period (from day 1 through day 29)
Description: A systematic adverse event is equivalent to an event that was solicited by the diary card, whereas a non-systematic event is equivalent to an event that was not solicited by the diary card.
Arm/Group | 2-10 Years | 11-18 Years | Overall (2 to 18 Years)
Serious Adverse Events (participants affected / at risk) | 1/173 | 0/167 | 1/340
Other Adverse Events (participants affected / at risk) | 110/173 | 98/167 | 208/340
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-10 Years (N=173) | 11-18 Years (N=167) | Overall (2 to 18 Years) (N=340)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 2-10 Years (N=173) | 11-18 Years (N=167) | Overall (2 to 18 Years) (N=340)
Nausea (Gastrointestinal disorders) | 10 (10) | 10 (10) | 20 (20)
Injection site erythema (General disorders) | 58 (58) | 43 (43) | 101 (101)
Injection site induration (General disorders) | 49 (49) | 36 (36) | 85 (85)
Injection site pain (General disorders) | 64 (64) | 62 (62) | 126 (126)
Malaise (General disorders) | 13 (13) | 35 (35) | 48 (48)
Nasopharyngitis (Infections and infestations) | 10 (10) | 2 (2) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 16 (16) | 6 (6) | 22 (22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 13 (13) | 16 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (20) | 49 (49) | 69 (69)
Headache (Nervous system disorders) | 13 (13) | 29 (29) | 42 (42)
Rash (Skin and subcutaneous tissue disorders) | 11 (11) | 4 (4) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No